CLINICAL TRIAL: NCT01448785
Title: Abiliti™ Treatment in Obese Subjects: A Randomized Post-Market Surveillance Multicenter Study
Brief Title: Abiliti™ Treatment in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IntraPace, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS-007-P
Record Dates: First submitted 2011-10-03; First posted 2011-10-07 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Obesity; Morbid Obesity
Keywords: obesity; gastric stimulation; morbid obesity
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- abiliti Group (Active Comparator): Subjects will receive implanted abiliti System. The device will be activated to deliver therapy at implant. Gastric stimulation performance testing, therapy adjustment and dietary/exercise counseling will be conducted at each visit.
  Interventions: Device: abiliti system implant
- Gastric Band Group (Active Comparator): Subjects will receive an implanted laparoscopic adjustable gastric band. The subjects will have their band adjusted following the standard of care. Dietary/exercise counseling will be conducted at each visit.
  Interventions: Device: Laparoscopic adjustable gastric band (Allergan Lap Band)

INTERVENTIONS:
Device: abiliti system implant — Subjects will receive implanted abiliti System.
  Other Names: abiliti
  Arms: abiliti Group
Device: Laparoscopic adjustable gastric band (Allergan Lap Band) — Subjects will receive an implanted laparoscopic adjustable gastric band. Specific brand is at the investigator's discretion.
  Other Names: gastric band
  Arms: Gastric Band Group

SUMMARY:
The main objective of this post-market surveillance study is to compare the subject's weight loss and quality of life, and device safety performance of the abiliti System and the adjustable gastric banding therapies in obese to morbidly obese subjects.

DETAILED DESCRIPTION:
This study is intended to provide additional data regarding the performance and safety of the abiliti system in comparison to gastric banding. The composite end-point of the study is designed to provide a direct comparison of the effectiveness of the devices for the treatment of obesity while giving consideration to the safety profile for each device and their impact on patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 60 years old at time of screening
* BMI of 40 to 55 or 35 to 39 with an obesity related comorbid condition at time of screening
* History of obesity ≥5 years
* The subject has been under routine care of the investigator or another single physician that can supply a medical record for at least 6 months prior to enrollment
* Women with childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods
* No significant weight loss (<5%) within four months prior to enrollment as documented in the subject's medical record.
* Successful psychological evaluation following the institution psychological evaluation protocol for bariatric surgery or successful historic assessment performed no more than 6 months prior to enrollment.
* Glycosylated Hemoglobin; HbA1c ≤ 7.0 % at Visit 2 or historic value performed no more than 3 months prior to enrollment.
* If taking anti-depressant medications, they must be stable for at least six months prior to enrollment
* Willingness to refrain from using prescription, over the counter or herbal weight loss products for the duration of the trial
* Alert, mentally competent, and able to understand and willing to comply with the requirements of the clinical trial, and personally motivated to abide by the requirements and restrictions of the clinical trial
* Able to provide voluntary informed consent

Exclusion Criteria:

* Any prior bariatric surgery
* Other implanted electrical stimulation devices (e.g. pacemaker, defibrillator, neurostimulator)
* Diagnosed with past or current psychiatric condition that may impair his/her ability to comply with the study procedures
* Use of anti-psychotic medications
* Diagnosed with a eating disorder such as bulimia or binge eating
* Obesity due to an endocrinopathy (e.g. Cushing disease)
* Insulin therapy
* GI disease such as hiatal hernia (>5cm), gastroparesis, esophageal motility disorders or intractable constipation.
* Cirrhosis, chronic pancreatitis
* History of intestinal obstruction or adhesive peritonitis
* Any history of peptic ulcer disease within 5 years prior to enrollment
* Women who are pregnant, lactating or anticipate becoming pregnant within 24 months
* Arthritis or other pathologies limiting physical activities that physician feels should exclude the patient from the study.
* Chronic use of aspirin and/or non steroidal anti-inflammatory medications and unwillingness to discontinue use
* Cardiac history that physician feels should exclude the patient from the study.
* Concurrent use of weight loss medications.
* Use of another investigational device or agent in the 30 days prior to enrollment
* A history of life-threatening disease within 5 years prior to enrollment
* Any other condition that, in the opinion of the investigator, would make the subject unsuitable for the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of the abiliti therapy compared to adjustable gastric banding | 12 months
  The non-inferiority of the abiliti therapy compared to adjustable gastric banding will be measured using a composite endpoint at the end of the study period. The success criteria will be the percentage of subjects in each group who meet all of the following criteria:
  * Achieve at least 20% excess weight loss (%EWL) from implant to end of the study period.
  * Experience no serious or severe adverse events related to the device or the procedure
  * No significant negative change in quality of life using the Impact Of Weight On Quality Of Life-Lite Questionnaire (IWQOL-Lite)
Percentage of Responders | 12 months
  Fifty (50 %) of the subject population must obtain an EWL ≥ 25%
Safety | 12 months
  * Incidence and seriousness of all adverse events.
  * Incidence of device or procedure-related adverse events
  * Frequency of clinically significant abnormal laboratory values as determined by the Investigator;

SECONDARY OUTCOMES:
Safety | 6 and 12 months
  Frequency of device and procedure-related adverse events
Quality of Life | 6 and 12 months
  Change in the quality of life using the IWQOL-Lite questionnaire
Eating Behavior | 6 and 12 months
  Change in the eating behavior (cognitive restraint, uncontrolled eating, and emotional eating) using the Three Factor Eating Questionnaire (TFEQ).
Co-morbid Conditions | 6 and 12 months
  Evaluation of the changes in blood pressure, lipid panel, HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Horbach, MD, Principal Investigator — Stadtkrankenhaus Schwabach; Alberic Fiennes, MD, Principal Investigator — St Anthony's Hospital, Surrey, England
Locations (15):
- Polyclinique de Rillieux, Clinique Lyon-Nord, Rillieux Cedex, France
- Germany (5):
  - MIC Ev. Krankenhaus Hubertus, Berlin
  - SRH Wald-Klinikum Gera, Gera
  - Wolfart Klinik, Gräfelfing
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Stadtkrankenhaus Schwabach, Schwabach
- Italy (3):
  - Azienda Ospedaliera- University, Pisa
  - Clinica San Luca Torino, Turin
  - Vicenza Regional Hospital, Vicenza
- Spain (2):
  - Complutense University of Madrid Hospital Clinico "San Carlos", Madrid
  - Hospital Virgen del Roció, Seville
- Klinik Lindberg, Winterthur, Switzerland
- United Kingdom (3):
  - Spire Southampton Hospital, Hampshire, Southampton
  - St. Anthony's Hospital, North Cheam, Surrey
  - Mid Yorkshire NHS Trust, Dewsbury, West Yorkshire

REFERENCES:
- [Derived] Morales-Conde S, Alarcon Del Agua I, Busetto L, Favretti F, Anselmino M, Rovera GM, Socas-Macias M, Barranco-Moreno A, Province-Azalde R, Torres AJ. Implanted Closed-Loop Gastric Electrical Stimulation (CLGES) System with Sensor-Based Feedback Safely Limits Weight Regain at 24 Months. Obes Surg. 2018 Jun;28(6):1766-1774. doi: 10.1007/s11695-017-3093-8. PMID 29333595
- [Derived] Busetto L, Torres AJ, Morales-Conde S, Alarcon Del Agua I, Moretto C, Fierabracci P, Rovera G, Segato G, Rubio MA, Favretti F. Impact of the feedback provided by a gastric electrical stimulation system on eating behavior and physical activity levels. Obesity (Silver Spring). 2017 Mar;25(3):514-521. doi: 10.1002/oby.21760. Epub 2017 Feb 6. PMID 28164463
- [Derived] Alarcon Del Agua I, Socas-Macias M, Busetto L, Torres-Garcia A, Barranco-Moreno A, Garcia de Luna PP, Morales-Conde S. Post-implant Analysis of Epidemiologic and Eating Behavior Data Related to Weight Loss Effectiveness in Obese Patients Treated with Gastric Electrical Stimulation. Obes Surg. 2017 Jun;27(6):1573-1580. doi: 10.1007/s11695-016-2495-3. PMID 28013450